CLINICAL TRIAL: NCT06270043
Title: A Prospective Registry and Longitudinal Study of Patients Undergoing Focal Therapy for Localized Prostate Cancer
Brief Title: Focal Therapy for Localized Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Juan Javier-DesLoges, Assistant Professor of Urology, University of California, San Diego
Other Study IDs: 809622
Record Dates: First submitted 2024-02-11; First posted 2024-02-21 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Focal Therapy; High Intensity Frequency Ultrasound; Transurethral Ultrasound Ablation; Cryoablation; Irreversible Electroporation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Urine and Blood samples will be collected on patients for bio banking and future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focal Therapy: Subjects who have biopsy-proven adenocarcinoma of the prostate, who have met all study inclusion and exclusion criteria, and have elected to receive or have already received focal therapy as part of their routine prostate cancer treatment, will be invited to participate in this observational registry study.
  Interventions: Procedure: Focal Therapy

INTERVENTIONS:
Procedure: Focal Therapy — Focal ablation of prostate cancer using different modalities. These modalities include:
  * Cryoablation or Cryotherapy
  * Irreversible Electroporation - Nanoknife
  * High Intensity Frequency Ultrasound - FocalOne
  * Transurethral Ultrasound Ablation - TULSA - PRO

SUMMARY:
This prospective registry and longitudinal study that is designed to carefully measure details of prostate cancer patients' outcomes with focal therapy. The goal of which is to improve patient care.

DETAILED DESCRIPTION:
This observational study will serve to collect data from medical record and review questionnaires before and after focal ablation of prostate tissue. All enrolled subjects will have already undergone or scheduled to receive the focal therapy as part of their prostate cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has elected or already undergone focal therapy as their standard of care treatment method and declined alternative treatment (active surveillance, radical prostatectomy, and radiation therapy)
* PSA ≤ 20
* Ability to complete informed consent form

Exclusion Criteria:

* Contraindication to follow-up multi parametric MRI or prostate biopsy
* Unable to tolerate general or regional anesthesia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Subjects who have biopsy-proven adenocarcinoma of the prostate, who have met all study inclusion and exclusion criteria, and have elected to receive or have already received the focal therapy as part of their routine prostate cancer treatment, will be invited to participate in this observational registry study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2034-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Oncological Response | 1 year
  The following definitions will be used for evaluation of oncological response:
  Complete response: Ablation of prostate tissue in targeted biopsy cores at 12 months.
  Incomplete response: Residual disease at 12 months compared to baseline in target biopsy cores or systematic biopsy cores.

SECONDARY OUTCOMES:
Erectile Dysfunction | 1 year
  Assess impact on erections after ablation. The Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) questionnaire will be used to evaluate sexual health quality-of-life symptoms for participants pre- and post-ablation.
  Patients will receive a score between 0 and 12, 0 being low with a better outcome and 12 being high with a worse outcome.
Incontinence | 1 year
  Assess impact on continence after ablation. The Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) questionnaire will be used to evaluate urinary health quality-of-life symptoms for participants pre- and post-ablation.
  Patients will receive a score between 0 and 12, 0 being low with a better outcome and 12 being high with a worse outcome.
Prostate cancer recurrence. Patients will be monitored with a Prostate Specific Antigen (PSA) every 6 months until 10 years from the intervention. Patients with a rising PSA will receive a prostate biopsy to determine if they have a recurrence. | 10 years
  Assess long-term recurrence risk after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Javier-DesLoges J, Dall'Era MA, Brisbane W, Chamie K, Washington SL 3rd, Chandrasekar T, Marks LS, Nguyen H, Daneshvar M, Gin G, Kane CJ, Bagrodia A, Cooperberg MR. The state of focal therapy in the treatment of prostate cancer: the university of California collaborative (UC-Squared) consensus statement. Prostate Cancer Prostatic Dis. 2024 Dec;27(4):579-581. doi: 10.1038/s41391-023-00702-1. Epub 2023 Aug 8. No abstract available. PMID 37553435